CLINICAL TRIAL: NCT01703260
Title: A Randomized, Double-Blind, Controlled, Multi-Center Phase 2 Study to Evaluate the Effect of Roflumilast Plus Pioglitazone on Liver Enzymes and Liver Fat Content in Subjects With Nonalcoholic SteatoHepatitis
Brief Title: Safety and Efficacy of Roflumilast and Pioglitazone in Treating Adults With Nonalcoholic SteatoHepatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision; No safety or efficacy concerns (see detailed description)
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ROF-NASH_205; U1111-1129-5051 (Registry Identifier: WHO)
Record Dates: First submitted 2012-10-02; First posted 2012-10-10 (Estimated); Results first posted 2016-02-23 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-09

CONDITIONS: Nonalcoholic Steatohapatitis
Keywords: Drug therapy
MeSH Terms: interventions — Roflumilast; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Roflumilast + pioglitazone (Experimental): Roflumilast dose and pioglitazone dose, orally for up to 4 months
  Interventions: Drug: Roflumilast; Drug: Pioglitazone
- Roflumilast (Experimental): Roflumilast dose and pioglitazone matching-placebo dose orally for up to 4 months.
  Interventions: Drug: Roflumilast; Drug: Placebo
- Pioglitazone (Experimental): Pioglitazone dose, orally and roflumilast matching-placebo dose, orally for up to 4 months
  Interventions: Drug: Pioglitazone; Drug: Placebo

INTERVENTIONS:
Drug: Roflumilast — Roflumilast dose
  Other Names: Daxas, Daliresp
  Arms: Roflumilast; Roflumilast + pioglitazone
Drug: Pioglitazone — Pioglitazone dose
  Other Names: Actos
  Arms: Pioglitazone; Roflumilast + pioglitazone
Drug: Placebo — Pioglitazone placebo-matching dose
  Arms: Roflumilast
Drug: Placebo — Roflumilast placebo-matching dose
  Arms: Pioglitazone

SUMMARY:
The purpose of this study is to evaluate the effect of roflumilast and pioglitazone therapy on serum transaminase (ALT) levels in adults with Nonalcoholic SteatoHepatitis.

DETAILED DESCRIPTION:
This proof of concept study will evaluate the effect of roflumilast and pioglitazone on transaminase levels and liver fat content.

Takeda has chosen not to continue this Study, however, randomized subjects were allowed to complete the study per protocol.

The decision to terminate the study is not related to any safety concerns with either of the study medications.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the patient is capable of understanding and complying with protocol requirements.
2. The patient or, when applicable, the patient's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Has a historical diagnosis of NASH, established no more than 12 months prior to study entry based on histology (liver biopsy).
4. Has a NAFLD Activity Score (NAS) of ≥3, with a score of at least 1 in steatosis and lobular inflammation - the subcomponents of NAS. It is acceptable if the score for hepatocyte ballooning is "zero".
5. The subject has a MRI determined liver fat fraction of equal or higher than 7 percent.
6. The subject is female or male and aged 18 to 80 years, inclusive.
7. A male who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 30 weeks after last dose.
8. A female of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study and for 30 days after last dose.
9. If taking Vitamin E and/or pentoxifylline, the subject has been receiving a stable dose for 6 months prior to randomization, started Vitamin E and/or pentoxifylline therapy prior to the qualifying liver biopsy, and agrees to maintain a stable dose throughout the study when possible.
10. Subject has an ALT level at Screening between 55 and 250 IU/L, inclusive, and between 60 and 250 IU/L at one other occasion during the 6 months prior to Randomization.
11. If taking a statin, should be on stable dose for 6 months prior to screening.
12. If taking angiotensin receptor blockers and fish oil, should be on a stable dose for at least 3 month prior to screening.
13. If diabetic, the subject is on a stable dose of metformin, dipeptidyl peptidase-4 inhibitor, sulfonylurea or insulin or a combination thereof for at least 3 months prior to Screening.

Exclusion Criteria:

1. The subject has a history of chronic liver disease other than NASH eg, chronic or acute hepatitis, Wilson's disease, alcoholic liver diseases or any other non-NASH active liver disease.
2. Subjects with liver cirrhosis (of any cause) or laboratory or clinical signs of functional liver failure
3. Clinically relevant abnormal laboratory values suggesting an undiagnosed disease other than NASH requiring further clinical evaluation (as assessed by the Investigator).
4. The subject has active cancer or a history of a malignant disease (except basal cell carcinoma) within 5 years prior to Screening or any history of bladder cancer.
5. Subject with a history of weight loss or weight gain of >10 pounds within 6 months prior to Screening.
6. Subject with a history of bariatric surgery within 5 years prior to Screening.
7. The subject has received any investigational compound within 30 days prior to Screening or is currently participating in another clinical study.
8. The subject has a history of hypersensitivity or allergies to roflumilast or pioglitazone including any associated excipients.
9. The subject is required to take excluded medications.
10. The subject has taken oral or injectable glucocorticoids for longer than 7 days within 3 months prior to Screening.
11. The subject has poorly controlled Type 1 or Type 2 diabetes mellitus with an HbA1c ≥8.5 at Screening or per Investigator judgment.
12. The subject has hepatitis A, B or C.
13. The subject has severe immunological diseases (eg, known HIV infection, multiple sclerosis, lupus erythematosus, progressive multifocal leukoencephalopathy) assessed at Screening.
14. The subject had a history of diabetic gastroparesis or history of gastric bypass surgery.
15. The subject had a history of coronary angioplasty, coronary stent placement, coronary bypass surgery, or myocardial infarction within 6 months prior to Screening.
16. The subject had New York Heart Association heart failure of Class (II-IV) regardless of therapy.
17. The subject had a diastolic blood pressure greater than 100 mm Hg or a systolic blood pressure of greater than 160 mm Hg (The mean of the 3 serial BP measurements will be used to determine subject eligibility).
18. The subject has presence or history of psychotic disorder that may be associated with suicidal thinking, ideation or behavior. These disorders include, but are not limited to, depression, psychosis, psychotic disorder, and schizophrenia. Subjects will be monitored by Columbia-Suicide Severity Rating Scales throughout the duration of the study.
19. The subject has a history of drug abuse (defined as illicit drug use) or a history of alcohol abuse (defined as regular or daily consumption of more than 2 alcoholic drinks per day for women or 3 alcoholic drinks per day for men. One drink is equivalent to a 12-ounce beer, a 4-ounce glass of wine, or a 1-ounce shot of hard liquor.) within 1 year prior to the Screening visit.
20. The subject has a hemoglobin <120 g/L for men and <100 g/L for women.
21. The subject has received pioglitazone or roflumilast in a previous clinical study or as a therapeutic agent within 1 year prior to screening.
22. If female, the subject is pregnant or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period.
23. The subject is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
24. The subject has significant results from physical examinations or clinical laboratory results that, at the discretion of the investigator, would make it difficult to successfully manage and follow the subject according to the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (3):
- United States (3):
  - Coronado, California
  - Annapolis, Maryland
  - Baltimore, Maryland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part at 11 sites in the United States from 26 April 2013 to 30 September 2014.
Pre-assignment Details: Participants with a historical diagnosis of nonalcoholic steatohepatitis (NASH) and nonalcoholic fatty liver disease (NAFLD) activity score (NAS) of greater than or equal to (>=) 3 were enrolled in 1 of 3 treatment groups as follows: roflumilast + pioglitazone; roflumilast only; pioglitazone only.
Groups:
- Roflumilast + Pioglitazone: Roflumilast, 500 microgram (mcg), tablet, orally, once daily and pioglitazone, 30 milligram (mg), tablet, orally, once daily for up to 4 months.
- Roflumilast Only: Roflumilast, 500 mcg, tablet, orally, once daily and pioglitazone placebo-matching tablet, orally, once daily for up to 4 months.
- Pioglitazone Only: Pioglitazone, 30 mg, tablet, orally, once daily and roflumilast placebo-matching tablet, orally, once daily for up to 4 months.
Period: Overall Study
Arm/Group | Roflumilast + Pioglitazone | Roflumilast Only | Pioglitazone Only
Started | 7 | 7 | 6
Completed | 4 | 3 | 3
Not Completed | 3 | 4 | 3
Not completed — Adverse Event | 1 | 2 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Study Termination | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The randomized set included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Roflumilast + Pioglitazone | Roflumilast Only | Pioglitazone Only | Total
Number analyzed (Participants) | 7 | 7 | 6 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (9.64) | 43.9 (14.77) | 42.5 (8.67) | 44.0 (10.93)
Age, Customized [Number; unit: participants]
  18 - 39 years | 3 | 2 | 3 | 8
  40 - 59 years | 4 | 4 | 3 | 11
  60 - 80 years | 0 | 1 | 0 | 1
Gender [Count of Participants; unit: Participants]
  Female | 5 | 2 | 2 | 9
  Male | 2 | 5 | 4 | 11
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 0 | 3 | 1 | 4
  Non-Hispanic or Latino | 7 | 4 | 5 | 16
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 2 | 0 | 2
  White | 7 | 4 | 6 | 17
  Multiracial | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 6 | 20
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 165.6 (15.13) | 168.7 (8.62) | 174.3 (7.50) | 169.3 (11.13)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 102.19 (21.041) | 92.06 (20.784) | 110.15 (15.456) | 101.03 (19.887)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter(kg/m^2)] | 37.18 (5.192) | 32.19 (6.189) | 36.60 (7.475) | 35.26 (6.381)
Smoking Classification [Number; unit: participants]
  Had Never Smoked | 3 | 6 | 5 | 14
  Current Smoker | 1 | 1 | 1 | 3
  Ex-Smoker | 3 | 0 | 0 | 3
Type 2 Diabetes Mellitus [Number; unit: participants]
  Had Diabetes Mellitus | 2 | 2 | 1 | 5
  Did Not Have Diabetes Mellitus | 5 | 5 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Amount of Serum Alanine Transaminase (ALT) at Baseline
Time Frame: Baseline
Population: Safety analysis set included all participants who were randomized, received at least 1 dose of double-blind study medication and had baseline assessment available.
Measure: Mean (Standard Deviation); unit: international units per liter (IU/L)
Arm/Group | Roflumilast + Pioglitazone | Roflumilast Only | Pioglitazone Only
Number analyzed (Participants) | 7 | 7 | 6
international units per liter (IU/L) | 101.7 (56.98) | 83.4 (31.63) | 118.8 (36.76)

2. Primary Outcome: Percent Change From Baseline in Serum ALT at Month 4
Description: The percent change between the serum ALT value collected at Month 4 or final visit relative to baseline.
Time Frame: Month 4
Population: Safety analysis set included all participants who were randomized, received at least 1 dose of double-blind study medication and had baseline and at least 1 post-baseline assessment available.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Roflumilast + Pioglitazone | Roflumilast Only | Pioglitazone Only
Number analyzed (Participants) | 3 | 3 | 3
percent change | -53.89 (23.362) | -56.22 (6.014) | -28.86 (53.298)

3. Secondary Outcome: Amount of Serum Aspartate Transaminase (AST) at Baseline
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Roflumilast + Pioglitazone | Roflumilast Only | Pioglitazone Only
Number analyzed (Participants) | 7 | 7 | 6
IU/L | 64.0 (43.49) | 44.9 (15.25) | 88.3 (73.06)

4. Secondary Outcome: Percent Change From Baseline in Serum AST at Month 4
Description: The percent change between the serum AST value collected at Month 4 or final visit relative to baseline.
Time Frame: Month 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Roflumilast + Pioglitazone | Roflumilast Only | Pioglitazone Only
Number analyzed (Participants) | 3 | 3 | 3
percent change | -41.31 (36.087) | -43.20 (7.339) | -17.56 (45.458)

5. Secondary Outcome: Liver Fat Content at Baseline
Description: Liver fat content was quantitatively measured by evaluating the percentage of proton density fat fraction (PDFF) from an abdominal magnetic resonance imaging (MRI). On the basis of Couinaud classification (a classification used to describe functional liver anatomy), the liver was divided into 8 segments: caudate, left superolateral, left inferolateral, left superomedial (4a), left inferomedial (4b), right anteroinferior, right posteroinferior, right posterosuperior and right anterosuperior.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of PDFF
Arm/Group | Roflumilast + Pioglitazone | Roflumilast Only | Pioglitazone Only
Number analyzed (Participants) | 7 | 7 | 6
percentage of PDFF
  Caudate; (n= 6, 7, 6) | 22.233 (8.2750) | 19.107 (7.7990) | 20.117 (9.8492)
  Left superolateral; (n= 6, 6, 6) | 19.485 (8.8080) | 17.813 (7.4410) | 17.278 (7.2225)
  Left inferolateral; (n= 6, 7, 6) | 22.385 (8.9894) | 19.747 (7.8306) | 19.153 (10.5909)
  Left superomedial: (n= 6, 7, 6) | 22.115 (9.7126) | 20.426 (7.9170) | 20.100 (9.8688)
  Left inferomedial: (n= 6, 6, 6) | 21.553 (9.5912) | 18.977 (8.6970) | 21.530 (9.5193)
  Right anteroinferior: (n= 6, 7, 6) | 22.478 (9.0548) | 19.994 (9.0103) | 20.742 (8.7829)
  Right posteroinferior: (n= 6, 7, 6) | 23.710 (8.6478) | 18.804 (6.6882) | 20.070 (9.9727)
  Right posterosuperior: (n= 6, 7, 6) | 23.282 (9.5984) | 18.870 (7.5764) | 19.943 (8.9666)
  Right anterosuperior: (n=6, 7, 6) | 23.630 (8.7454) | 19.786 (8.5929) | 21.527 (9.6648)

6. Secondary Outcome: Change From Baseline in Liver Fat Content at Month 4
Description: Liver fat content was quantitatively measured by evaluating the percentage of PDFF from an abdominal MRI. On the basis of Couinaud classification (a classification used to describe functional liver anatomy), the liver was divided into 8 segments: caudate, left superolateral, left inferolateral, left superomedial (4a), left inferomedial (4b), right anteroinferior, right posteroinferior, right posterosuperior and right anterosuperior.
Time Frame: Baseline and Month 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change in PDFF
Arm/Group | Roflumilast + Pioglitazone | Roflumilast Only | Pioglitazone Only
Number analyzed (Participants) | 7 | 7 | 6
percent change in PDFF
  Caudate; (n= 3, 3, 3) | -18.787 (11.5646) | -11.590 (5.5674) | -10.287 (8.8098)
  Left superolateral; (n= 6, 6, 6) | -15.170 (13.7442) | -10.287 (1.9695) | -8.067 (7.6318)
  Left inferolateral; (n= 3, 3, 3) | -14.290 (13.1654) | -10.077 (2.9030) | -8.773 (7.0821)
  Left superomedial: (n= 3, 3, 3) | -14.687 (13.6909) | -11.177 (3.9429) | -9.217 (8.7999)
  Left inferomedial: (n= 3, 3, 3) | -14.107 (15.2957) | -10.977 (5.0052) | -9.417 (8.9360)
  Right anteroinferior: (n= 3, 3, 3) | -13.990 (13.1266) | -10.260 (6.9972) | -7.693 (9.7985)
  Right posteroinferior: (n=3, 3, 3) | -18.073 (13.1470) | -9.250 (1.6808) | -8.790 (10.2188)
  Right posterosuperior: (n=3, 3, 3) | -17.717 (13.0691) | -9.797 (4.4053) | -8.113 (10.4166)
  Right anterosuperior: (n=3, 3, 3) | -16.127 (13.9820) | -9.803 (3.3661) | -8.647 (10.1658)

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs will be defined as any AEs, regardless of relationship to study drug, that occur or worsen after the first dose of double-blinded study drug and no more than 30 days after the last dose of study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Roflumilast + Pioglitazone | Roflumilast Only | Pioglitazone Only
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 5/7 | 4/7 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Roflumilast + Pioglitazone (N=7) | Roflumilast Only (N=7) | Pioglitazone Only (N=6)
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 2
Weight decreased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0
Cow's milk intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.